CLINICAL TRIAL: NCT04110509
Title: Fragility and Programmed Cardiovascular Surgery: Development of Muscle Ultrasonographic Biomarkers of Sarcopenia and Post-surgical Results
Brief Title: Fragility and Programmed Cardiovascular Surgery (EcoSarco)
Acronym: EcoSarco
Status: Completed | Type: Observational
Sponsor: Universidad Antonio de Nebrija (Other)
Responsible Party: Principal Investigator, José Ríos-Díaz, PhD in Biology, Physical Therapist, Universidad Antonio de Nebrija
Other Study IDs: ECOSARCO_CARDIO v0.2
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Fragility; Intensive Care Unit Syndrome
Keywords: Imaging biomarkers; Ultrasonography; Fragility; Intensive Care Unit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives: To characterize textural ultrasonographic biomarkers of the brachial biceps musculature, wrist flexors, quadriceps and anterior tibial muscle that allow the recognition of the muscular and functional status of patients undergoing programmed cardiovascular surgery and relate them to mortality, hospital stay and functionality results after the intervention.

Design: A first phase of cross-sectional observational study and a second phase of longitudinal observational prospective study. Participants: Patients with programmed cardiovascular surgery to aortic valve replacement Outcomes: Sociodemographic and anthropometric variables, severity and clinical risk scales, disability, fragility and quality of life scales, nutritional status and textural muscular biomarkers with ultrasonography.

Expected results: strong association between ultrasound muscle biomarkers and ICU and hospital stay, disability, fragility and quality of life after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Waiting list patients with cardiovascular surgery scheduled for aortic valve refill

Exclusion Criteria:

* Urgency while waiting list
* Patients with no evaluation by presurgery committee
* Previous diagnosis of neuropathies, radiculopathy, polyneuropathy congenital or acquired or pathologies with muscular affectation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the Intensive Care Unit of the Hospital Clínico Universitario Virgen de la Arrixaca de Murcia (HCUVAM) and the Hospital Universitario del Vinalopó de Elche (HUVE) for surgery programmed cardiovascular, specifically aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in muscle ultrasonography variation after surgery | 6 months
  Ultrasonography variation is a measure of the degree of heterogeneity of a ultrasonographic image which provides information on changes in tissue structure (muscles).
Changes in muscle echointensity after surgery | 6 months
  Echointensity is the average of echogenicity of a ultrasonographic image which provides information on changes in tissue structure
Changes in muscle texture after surgery | 6 months
  Muscle texture can be characterized by advanced image analysis algorithms such grey level co-occurrence matrices. In this case 5 textural parameters (uniformity, contrast, homogeneity, correlation and entropy) used together are used to characterize the tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Rios-Diaz, Madrid, Spain